CLINICAL TRIAL: NCT02126150
Title: United CORoNary Biobanks
Acronym: UNICORN
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Crystel Gijsberts, MD, UMC Utrecht
Other Study IDs: 11-183
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Stable Angina
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, peripheral blood mononuclear cells and whole blood is stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ethnicity

SUMMARY:
The UNICORN consists of two collaborating biobanks, one in Utrecht and one in Singapore. From these two sites we include all patients who undergo a coronary catheterization for any reason.

At the moment of catheterization we draw blood, which will be stored in a biobank and we collect clinical characteristics. Patients are followed-up for 5 years for the occurrence of major cardiovascular events.

By including from two sites in the world we include 4 major ethnic groups: Caucasians, Chinese, Indians and Malays. We aim at including at least 2000 patients per ethnic group.

Our hypothesis is that there are differences in the risk factor burden, clinical presentation of CAD, and biochemical patterns in the blood among the ethnic groups.

Furthermore, this biobank offers a platform for multi-ethnic biomarker discovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography

Exclusion Criteria:

* < 21 years of age
* Hemoglobin levels <7 g/dL in women, or hemoglobin levels <8 g/dL in men

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that undergo coronary catheterization for any reason are eligible to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
All-cause death | 5 years

SECONDARY OUTCOMES:
Major cardiovascular events | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore